CLINICAL TRIAL: NCT04623541
Title: A Phase 1b/2, Open-Label, Safety and Efficacy Study of Epcoritamab (GEN3013; DuoBody®-CD3xCD20) in Relapsed/Refractory Chronic Lymphocytic Leukemia and Richter's Syndrome
Brief Title: Safety and Efficacy Study of Epcoritamab in Subjects With Relapsed/Refractory Chronic Lymphocytic Leukemia and Richter's Syndrome
Acronym: EPCORE™ CLL-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT3013-03; 2020-000848-57 (EudraCT Number); NL74221.056.20 (Registry Identifier: CCMO); MOH_2023-04-02_012496 (Registry Identifier: MyTrial); 2023-504828-25-00 (EU CTIS Number); 1006575 (Other: IRAS ID; UK Research Summaries Database); RECF-005228 (Other: Nationale Institute of Cancer Research)
Expanded Access: NCT05733650 (Approved for marketing)
Record Dates: First submitted 2020-10-27; First posted 2020-11-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Relapsed/Refractory Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Richter's Syndrome; Treatment-naïve High Risk Chronic Lymphocytic Leukemia
Keywords: DuoBody®; Bispecific antibodies; Anti-CD3; Anti-CD20
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; venetoclax; Lenalidomide; pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Epcoritamab in R/R CLL/SLL (Experimental): In both study phases. Participants in the expansion phase will be treated at the RP2D defined in the dose-escalation phase.
  Interventions: Biological: Epcoritamab
- Epcoritamab in RS (Experimental): Only in expansion phase.
  Interventions: Biological: Epcoritamab
- Epcoritamab + Venetoclax in R/R CLL/SLL (Experimental): In both study phases. Participants in the expansion phase will be treated at the RP2D defined in the dose-escalation phase.
  Interventions: Biological: Epcoritamab; Drug: Venetoclax
- Epcoritamab + Lenalidomide in RS (Experimental): Only in expansion phase.
  Interventions: Biological: Epcoritamab; Drug: Lenalidomide
- Epcoritamab + R-CHOP in RS (Experimental): Only in expansion phase.
  Interventions: Biological: Epcoritamab; Drug: rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone
- Epcoritamab + Pirtobrutinib in R/R CLL, TN HR CLL (Non-US Participants Only) and SLL (Experimental): Safety run-in and expansion phases.
  Interventions: Biological: Epcoritamab; Drug: Pirtobrutinib
- Fixed Duration Epcoritamab in R/R CLL/SLL (Experimental): Only in expansion phase.
  Interventions: Biological: Epcoritamab

INTERVENTIONS:
Biological: Epcoritamab — Epcoritamab will be administered subcutaneously in cycles of 28 days, (except Cycle 1 for high-dose cohorts = 35 days).
  Other Names: EPKINLY™; GEN3013; DuoBody®-CD3xCD20
  Arms: Epcoritamab + Venetoclax in R/R CLL/SLL; Epcoritamab in R/R CLL/SLL
Biological: Epcoritamab — Epcoritamab will be administered subcutaneously in cycles of 21 days and 28 days.
  Other Names: EPKINLY™; GEN3013; DuoBody®-CD3xCD20
  Arms: Epcoritamab + R-CHOP in RS
Drug: rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone — R-CHOP will be administered intravenously (prednisone may be administered orally) in cycles of 21 days.
  Arms: Epcoritamab + R-CHOP in RS
Drug: Venetoclax — Venetoclax tablets will be administered orally once daily during the 5-week ramp up period in cycles of 28 or 35 days each.
  Arms: Epcoritamab + Venetoclax in R/R CLL/SLL
Biological: Epcoritamab — Epcoritamab will be administered subcutaneously in cycles of 28 days.
  Other Names: EPKINLY™; GEN3013; DuoBody®-CD3xCD20
  Arms: Epcoritamab + Lenalidomide in RS; Epcoritamab in RS
Drug: Lenalidomide — Lenalidomide capsules will be administered once daily for 21 days in each cycle of 28 days.
  Arms: Epcoritamab + Lenalidomide in RS
Biological: Epcoritamab — Epcoritamab will be administered subcutaneously in cycles of 28 days.
  Other Names: EPKINLY™; GEN3013; DuoBody®-CD3xCD20
  Arms: Epcoritamab + Pirtobrutinib in R/R CLL, TN HR CLL (Non-US Participants Only) and SLL
Drug: Pirtobrutinib — Pirtobrutinib tablets will be administered in cycles of 28 days.
  Arms: Epcoritamab + Pirtobrutinib in R/R CLL, TN HR CLL (Non-US Participants Only) and SLL
Biological: Epcoritamab — Epcoritamab will be administered subcutaneously in cycles of 28 days.
  Other Names: EPKINLY™; GEN3013; DuoBody®-CD3xCD20
  Arms: Fixed Duration Epcoritamab in R/R CLL/SLL

SUMMARY:
The study is a global, multi-center safety and efficacy trial of epcoritamab, an antibody also known as EPKINLY™ and GEN3013 (DuoBody®-CD3xCD20). Epcoritamab will be tested either in

Relapsed/refractory (R/R) chronic lymphocytic leukemia (CLL) as:

* Monotherapy, or
* Combination therapy:

  * epcoritamab + venetoclax
  * epcoritamab + pirtobrutinib

In Non-United States (US) Participants Only: Treatment-naïve (TN) high risk (HR) (CLL):

• epcoritamab + pirtobrutinib

Combination therapy for Richter's Syndrome (RS):

* epcoritamab + lenalidomide
* epcoritamab + R-CHOP (i.e., rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine [Oncovin®] and prednisone).

The study includes participants with R/R or TN HR CLL (non-US participants only)/small lymphocytic lymphoma (SLL) and participants with RS.

The trial consists of two parts, a dose-escalation phase (phase Ib) and an expansion phase (phase II). Participants with RS are only included in the expansion phase.

Epcoritamab will be injected subcutaneously (under the skin). Standard-of-care and combination treatments (venetoclax, pirtobrutinib, lenalidomide, and R-CHOP) will be given either orally (by mouth) or intravenously (in a vein).

Study details include:

* Study duration will be up to 5 years after the last participant's first treatment in the trial.
* The treatment duration for each participant will be between 12 months (1 year) and 24 months (2 years), depending upon the treatment arm assigned.
* The visit frequency will be either weekly, every other week, or monthly, depending upon the part of the study.

All participants will receive active drug; no one will be given placebo.

DETAILED DESCRIPTION:
The purpose of the dose-escalation phase of the trial is to determine the recommended phase 2 dose (RP2D) and the maximum tolerated dose (MTD; if reached) as well as establish the safety profile of epcoritamab monotherapy and epcoritamab + venetoclax in participants with R/R CLL.

The purpose of the expansion phase is to assess and evaluate the preliminary efficacy, safety and tolerability profiles of epcoritamab monotherapy, epcoritamab + venetoclax and epcoritamab + pirtobrutinib at the RP2D for participants with R/R CLL, TN HR CLL (in non-US participants only) and SLL. Along with this, epcoritamab monotherapy, epcoritamab + lenalidomide and epcoritamab + R-CHOP will be evaluated in participants with RS to assess their efficacy, safety and tolerability profiles.

The purpose of safety run-in phase for pirtobrutinib combination therapy is to evaluate the safety and tolerability profiles of pirtobrutinib in combination with epcoritamab.

ELIGIBILITY:
Key Inclusion Criteria

1. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2.
2. Evidence of CD20 positivity in a sample representative of the disease at Screening.
3. Acceptable hematology parameters and organ function based on baseline bloodwork.
4. Life expectancy >3 months on standard of care (SOC) for CLL, >3 months for RS.
5. For R/R CLL arms - Must have active CLL/SLL disease requiring treatment per iwCLL 2018 criteria.
6. For R/R CLL monotherapy arms - Received at least 2 prior lines of systemic anti-neoplastic therapy including a Bruton's tyrosine kinase (BTK) inhibitor or at least 1 prior line of systemic antineoplastic therapy, including treatment with (or intolerance of) a covalent BTK inhibitor (cBTKi) and a B-cell lymphoma 2 (BCL-2) inhibitor.
7. For all RS arms - Have tumor biopsy-proven CD20+ Diffuse large B-cell Lymphoma (DLBCL) and a clinical history of CLL/SLL.
8. For all RS arms - Must have measurable disease by fluorodeoxyglucose-positron emission tomography (FDG-PET) and computed tomography (CT) or magnetic resonance imaging (MRI) scan.
9. For all RS arms - Must provide mandatory formalin-fixed, paraffin-embedded (FFPE) tumor biopsy sample.
10. For RS - monotherapy arm: Deemed as ineligible for chemoimmunotherapy at investigator's discretion or participant who refuses to receive intensive chemotherapy
11. For RS - lenalidomide combination therapy arm

    * Deemed as ineligible for chemoimmunotherapy at the investigator's discretion, or participant who refuses to receive intensive chemotherapy.
    * Eligible for treatment with lenalidomide.
    * Must be willing to use contraception and adhere to the Lenalidomide Pregnancy Risk Minimization Plan
    * A woman must agree not to breastfeed a child during treatment and for at least 28 days after discontinuation from study.
12. For RS - R-CHOP combination Therapy Arm -

    * Eligible for treatment with R-CHOP.
    * Females of childbearing potential must use highly effective contraceptive measures while taking R-CHOP and for 12 months after stopping treatment.
    * A woman must agree not to breastfeed a child during treatment or until 12 months after last treatment.
13. For R/R CLL - venetoclax combination Therapy arm - after receiving at least 1 prior line of systemic antineoplastic therapy.

    * Presence of measurable disease.
    * Must take prophylaxis for tumor lysis syndrome (TLS).
14. For R/R CLL pirtobrutinib combination Therapy arm:

    * Must have active CLL/SLL disease requiring treatment per iwCLL 2018 criteria.
    * Presence of measurable disease.
    * Previous treatment with at least one and a maximum 3 prior lines of therapy including a cBTKi.
    * Diagnosis of CLL/SLL that met published iwCLL criteria.
15. Non-US Participants Only - Participants with TN HR CLL - Pirtobrutinib Combination Therapy Expansion:

    * Diagnosis of CLL/SLL that met published iwCLL criteria 2018.
    * Must have active CLL/SLL disease that needs treatment per iwCLL
    * Must take prophylaxis for TLS based on their TLS risk evaluation upon initiation of trial drug.
    * Must have one or more high-risk features.
    * Presence of measurable disease.

Key Exclusion Criteria

1. Received prior treatment with a CD3×CD20 bispecific antibody.
2. Received any prior allogeneic hematopoietic stem cell transplantation (HSCT) or solid organ transplantation.
3. Received chimeric antigen receptor (CAR) T-cell therapy within 100 days or an investigational drug within 4 weeks, prior to first dose of trial drug.
4. Autoimmune disease or other diseases that require permanent or high-dose immunosuppressive therapy.
5. Received vaccination with live vaccines within 28 days.
6. Clinically significant cardiac disease.
7. Known current malignancy other than inclusion diagnosis.
8. Has had major surgery within 4 weeks.
9. Known history of human immunodeficiency virus (HIV).
10. For R/R CLL arms - Any history of RS or evidence indicating a potential Richter's transformation.
11. For R/R CLL - Venetoclax Combination Therapy arm: received venetoclax within 24 months prior to beginning venetoclax ramp-up for this trial or has progressed on venetoclax treatment.
12. For all RS arms - Diagnosis of Richter's syndrome not of the DLBCL subtype such as Hodgkin's lymphoma, prolymphocytic leukemia.
13. RS - Lenalidomide Combination Therapy and RS Monotherapy Arms - received more than 2 prior lines of therapy for RS.
14. R/R CLL - Pirtobrutinib Combination Therapy Arm - Prior exposure to a non-covalent (reversible) BTK inhibitor or a BTK degrader.
15. Pirtobrutinib Combination Therapy Expansion Arms:

    * History of bleeding disorders or participants requiring therapeutic anticoagulation with warfarin or another vitamin K antagonist
    * Require continuous treatment with or have received strong cytochrome P450 (CYP) 3A inhibitors or strong/moderate CYP3A inducers within 4 to 5 half-lives or 14 days prior to the first dose of pirtobrutinib.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Phase and Safety Run-in (R/R CLL arm): Number of Participants with Dose Limiting Toxicities (DLTs) | During the first cycle for low dose cohorts (Cycle length = 28 days) and for high dose cohorts (Cycle length = 35 days)
  DLT events were defined as clinically significant adverse events (AEs) or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications as assessed per Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0.
Dose Escalation Phase and Safety Run-in: Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 5 years
Dose Escalation Phase: Number of Participants with Cytokine Release Syndrome (CRS), Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) and Clinical Tumor Lysis Syndrome (CTLS) | Up to 5 years
  CRS and ICANS will be graded based on American Society for Transplantation and Cellular Therapy (ASTCT) criteria. CTLS will be graded according to Cairo-Bishop criteria.
Expansion Phase: Overall Response Rate (ORR) | Up to 5 years
  R/R CLL participants will be assessed according to International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria and the RS participants according to Lugano criteria. ORR based on the Lugano criteria is defined as the percentage of participants who achieve a response of PR or complete remission (CR), prior to initiation of subsequent therapy. The ORR based on the iwCLL criteria is defined as the percentage of participants who achieve a response of PR, CR with incomplete bone marrow recovery (CRi), or CR, prior to the initiation of subsequent therapy.

SECONDARY OUTCOMES:
Expansion Phase: Number of Participants with TEAEs and SAEs | Up to 5 years
Dose Escalation Phase and Safety Run-in: ORR (for R/R CLL Participants) | Up to 5 years
  The ORR is defined as the percentage of participants who achieve a response of PR, CRi, or CR, prior to the initiation of subsequent therapy as assessed by iwCLL criteria.
Both Phases and Safety Run-in: Duration of Response (DOR) | Up to 5 years
  DOR is defined among responders, as the time from the initial documentation of response to the date of disease progression or death, whichever occurs earlier.
Both Phases and Safety Run-in: Number of Participants with CR/CRi | Up to 5 years
  CR and CRi for R/R CLL participants will be assessed according to iwCLL criteria and CR for the RS participants, according to Lugano criteria.
Both Phases and Safety Run-in: Time to Response (TTR) | Up to 5 years
  TTR is defined among responders, as the time between first dose of any study drug and the initial documentation of response.
Both Phases and Safety Run-in: Progression Free Survival (PFS) | Up to 5 years
  PFS is defined as the time from the first dosing date of any study drug and the date of disease progression or death, whichever occurs earlier.
Both Phases and Safety Run-in: Overall Survival (OS) | Up to 5 years
  OS is defined as the time from the first dosing date of any study drug and the date of death due to any cause.
Both Phase and Safety Run-in: Time to Next Systemic Anti-cancer Therapy (TTNT) | Up to 5 years
  TTNT is defined as the time from the first dosing date of any study drug to the first documented administration of subsequent systemic anticancer therapy.
Both Phases and Safety Run-in: Area Under the Concentration-time Curve (AUC) in Epcoritamab | Predose and post dose at multiple timepoints at end of each cycle for low dose and high dose cohorts (Cycle length = 28 days, except Cycle 1 for high dose cohorts = 35 Days), up to 5 years
Both Phases and Safety Run-in: Maximum (Peak) Plasma Concentration (Cmax) in Epcoritamab | Predose and post dose at multiple timepoints at end of each cycle for low dose and high dose cohorts (Cycle length = 28 days, except Cycle 1 for high dose cohorts = 35 Days), up to 5 years
Both Phases: Pre-dose (Trough) Concentrations (Cthrough) in Epcoritamab | Predose and post dose at multiple timepoints at end of each cycle for low dose and high dose cohorts (Cycle length = 28 days, except Cycle 1 for high dose cohorts = 35 Days), up to 5 years
Both Phases and Safety Run-in: Time to Reach Cmax (Tmax) in Epcoritamab | Predose and post dose at multiple timepoints at end of each cycle for low dose and high dose cohorts (Cycle length = 28 days, except Cycle 1 for high dose cohorts = 35 Days), up to 5 years
Both Phases and Safety Run-in: Elimination Half-life (T1/2) in Epcoritamab | Predose and post dose at multiple timepoints at end of each cycle for low dose and high dose cohorts (Cycle length = 28 days, except Cycle 1 for high dose cohorts = 35 Days), up to 5 years
Both Phases and Safety Run-in: Total Body Clearance of Drug From Plasma (CL) in Epcoritamab | Predose and post dose at multiple timepoints at end of each cycle for low dose and high dose cohorts (Cycle length = 28 days, except Cycle 1 for high dose cohorts = 35 Days), up to 5 years
Both Phases: Lymphoid Cells for Immunophenotyping | Up to 5 years
  Evaluation of B cells, T cells and their activation
Expansion Phase: Number of Participants with CRS, ICANS and CTLS | Up to 5 years
  CRS and ICANS will be graded based on ASTCT criteria. CTLS will be graded according to Cairo-Bishop criteria.
Expansion Phase and Safety Run-in : Percentage of Participants with Minimal Residual Disease (MRD) Negativity | Up to 5 years
  MRD negativity rate, is defined as the proportion of participants with at least 1 undetectable MRD result according to the specific threshold, prior to initiation of subsequent therapy.
Both Phases and Safety Run-in: Number of Participants with Anti-drug Antibodies (ADA) to Epcoritamab | Up to 5 years
Expansion Phase: Number of Participants with PR | Up to 5 years
Both Phases and Safety Run-in: Duration of MRD Negativity | Up to 5 years
  The time from first achieving MRD negativity after start of treatment to the MRD conversion to positive.

CONTACTS AND LOCATIONS:
Locations (87):
- United States (23):
  - O'Neal Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Davis Medical Center Sacramento, California City, California
  - City of Hope National Medical Center, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - David Geffen School of Medicine, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - National Institutes of Health, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Medical Group, Detroit, Michigan
  - Hackensack Meridian Hospital, Hackensack, New Jersey
  - Northwell Health Cancer Institute, Lake Success, New York
  - Columbia University Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania School of medicine, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Centre, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (5):
  - St. George Hospital, Kogarah, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Barwon Health, Geelong, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria
- Belgium (3):
  - AZ Sint-Jan, Bruges
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Czechia (5):
  - Vseobecna Fakultni Nemocnice, Prague, Nové Město
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Nový Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava, Poruba
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
- Denmark (6):
  - Rigshospitalet, Copenhagen, Capital Region
  - Aalborg University Hospital, Aalborg
  - Århus University Hospital, Aarhus
  - Odense University Hospital, Odense
  - Roskilde Sygehus, Roskilde
  - Vejle Sygehus, Vejle
- France (7):
  - CHU de Montpellier Hôpital Saint Eloi, Montpellier, Cedex 5
  - CHU Hôpital Haut-Lévêque Bordeaux, Pessac, Gironde
  - CHU Hôpital de Brabois Nancy, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Hôpital Privé du Confluent, Nantes, Pays de la Loire Region
  - CHU Clermont Ferrand, Clermont-Ferrand, Puy De Dome
  - Hôpital Saint-Louis, Paris
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
- Germany (3):
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Schleswig-Holstein- Karl-Lennart-Krebscentrum, Kiel
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - Istituto di Candiolo, Torino, Candiolo
  - AOU Arcispedale Sant'Anna, Ferrara, Cona
  - IRCCS Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori IRST, Meldola, Forli - Cesena
  - IRCCS Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - AOU Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Ospedale San Raffaele, Milan
  - Ospedale Maggiore di Novara, Novara
  - AOU Policlinico Umberto I, Roma
  - AOU Città della Salute e della Scienza di Torino, Torino
- Netherlands (5):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Albert Schweitzer Ziekenhuis, Dordwijk, Dordrecht, South Holland
  - Amsterdam UMC, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (3):
  - Pratia Medical Center Katowice (Centrum Medyczne Pratia Katowice), Katowice
  - Pratia Malopolskie Medical Center Krakow (Pratia Małopolskie Centrum Medyczne Krakow), Krakow
  - Aidport sp z o.o., Skorzewo
- Spain (8):
  - ICO Badalona - Hospital Universitario Germans Trias Pujol, Badalona, Barcelona
  - AOC Arcispedale Saint'Anna, Coaña, Ferarra
  - Hospital Clinico Universitario de Valencia, Valencia, València
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundacion Jiménez Díaz, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (4):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Nottingham University Hospitals City Campus, Nottingham, Nottinghamshire
  - St. James s University Hospital, Leeds, West Yorkshire
  - Barts Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kater AP, Janssens A, Eradat H, Offner F, Sandoval-Sus JD, Shadman M, Poulsen CB, Christensen JH, Thompson MC, Guan M, Steele AJ, Rios M, Holst Morch M, Oki T, Valentin R, Bellido M, Eichhorst B. Epcoritamab monotherapy for Richter transformation (EPCORE CLL-1): findings from a single-arm, multicentre, open-label, phase 1b/2 trial. Lancet Haematol. 2026 Jan;13(1):e8-e21. doi: 10.1016/S2352-3026(25)00327-8. Epub 2025 Dec 8. PMID 41380698